CLINICAL TRIAL: NCT06135779
Title: Evaluation of the Effectiveness of a Universal School-based Intervention to Improve the Well-being of Children Aged 8-11 Years.
Brief Title: Evaluation of the Effectiveness of a School-based Intervention to Improve the Wellbeing of Children Aged 8-11 Years.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-22-80-Carr
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Well-Being, Psychological; Child, Only
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Lust for Life programme group (Experimental): A Lust for Life programme will be delivered to participants by their class teachers in ten weekly sessions
  Interventions: Behavioral: A Lust for Life
- Waiting list control group (Other): Participants will receive curriculum as usual from their class teacher, and placed on a 12-week waiting list for the programme.
  Interventions: Behavioral: Waiting List Control

INTERVENTIONS:
Behavioral: A Lust for Life — A Lust For Life (ALFL) is a universal teacher-led programme which aims to build resilience, increase wellbeing, and enhance emotional literacy of 8-13 year old school children. The programme spans ten 40-minute classes. The ALFL curriculum draws on multiple sources including contemporary positive psychology; traditional, second, and third wave cognitive behaviour therapy (CBT); and developmental, educational, and health psychology. In ALFL children learn the following specific self-regulation skills: naming and rating the intensity of emotions; linking thoughts, feelings and actions; mindfulness; breathing exercises; visualization exercises; progressive muscle relaxation; positive self-talk (gratitude, optimism, and cognitive restructuring); obtaining social support from adults and peers; assertiveness; managing bullying; and using the internet safely. Skills are learned through didactic instruction, video modelling, in-class experiential exercises, and homework practice.
  Arms: A Lust for Life programme group
Behavioral: Waiting List Control — Control group placed on a 12-week waiting list for the A Lust for Life School programme.
  Arms: Waiting list control group

SUMMARY:
The aim of this study is to evaluate the effectiveness of a universal school-based intervention, which aims to improve the wellbeing of children aged 8 to 11 years, who are attending 3rd class or 4th class in primary level education in Ireland.

DETAILED DESCRIPTION:
An estimated 10-20% of children and adolescents worldwide experience mental health difficulties, with 50% of difficulties emerging before the age of 14 years. School is an influential environment for young people, with school-based interventions consistently delivering positive mental health and wellbeing programmes in a cost-effective manner.

A Lust for Life (ALFL) is a universal teacher-led programme which aims to build resilience, increase wellbeing, and enhance emotional literacy of 8-13 year old school children. The programme spans ten 40-minute classes. The ALFL curriculum draws on multiple sources including contemporary positive psychology; traditional, second, and third wave cognitive behaviour therapy (CBT); and developmental, educational, and health psychology. In ALFL children learn the following specific self-regulation skills: naming and rating the intensity of emotions; linking thoughts, feelings and actions; mindfulness; breathing exercises; visualization exercises; progressive muscle relaxation; positive self-talk (gratitude, optimism, and cognitive restructuring); obtaining social support from adults and peers; assertiveness; managing bullying; and using the internet safely. Skills are learned through didactic instruction, video modelling, in-class experiential exercises, and homework practice. The ongoing development of the ALFL programme follows best practice, with the most recently refined programme evaluated in this study.

This quasi-experimental randomized controlled trial study involves an experimental group and a waiting list control group of children aged between 8-11 years. All study participants will complete the Feeling Better Scale, Stirling Children's Wellbeing Scale, and Revised Children's Anxiety and Depression Scale at pre-intervention. Participants will complete the questionnaires online. Following this, schools randomly assigned to the experimental group will receive the ALFL programme, while those randomly assigned to the control group will be placed on a 12-week waiting list and receive curriculum as usual. At post-intervention, the questionnaire measures will be completed online by all study participants. The participants in the experimental group will also complete a brief Satisfaction Scale. The waiting list control group will then receive the A Lust for Life programme.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-11 years
* Enrolled in 3rd and 4th classes in Primary School in Ireland
* Obtain written informed consent from parents/guardians
* Provide written assent

Exclusion Criteria:

* Failure to meet inclusion criteria

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Wellbeing measured by the Feeling Better Scale | 10 weeks after beginning the intervention
  Scores on the Feeling Better Scale range from 0 to 152. Higher scores indicate higher levels of wellbeing.

SECONDARY OUTCOMES:
Wellbeing measured by the Stirling Children's Wellbeing Scale | 10 weeks after beginning the intervention
  Scores on the Stirling Children's Wellbeing Scale range from 12 to 60. Higher scores indicate higher wellbeing.
Anxiety and low mood measured by the Revised Children's Anxiety and Depression Scale | 10 weeks after beginning the intervention
  Scores on the Revised Children's Anxiety and Depression Scale range from 0 to 75. Higher scores indicate greater severity of anxiety and low mood.
Programme Satisfaction with the Satisfaction Scale | 10 weeks after beginning the intervention
  Scores on the Satisfaction Scale range from 8 to 56. Higher scores indicate higher satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Alan Carr, Professor, Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data collected in this research will be archived. Other researchers may contact the investigators to access the de-identified data for use in research into well-being.
Supporting Information: Study Protocol
Time Frame: The data collected in this study will be made available for other researchers after a manuscript reporting on the study's findings has been accepted for publication.
Access Criteria: Data may be accessed for use in research into well-being.